CLINICAL TRIAL: NCT02793830
Title: A Mobile Phone Based Medication Reminder Program for Patients in China With Coronary Heart Disease: A Pilot Study
Brief Title: A Mobile Phone Based Medication Reminder Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00073395
Record Dates: First submitted 2016-06-03; First posted 2016-06-08 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Medication Adherence
Keywords: medication adherence; mHealth; China; heart disease
MeSH Terms: conditions — Medication Adherence; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mobile App Group (Experimental): Participants in the experimental group will receive daily reminders and educational materials from mobile applications.
  Interventions: Other: Daily reminders of taking medications; Other: Educational materials
- Control Group (Active Comparator): The control group will receive the same educational materials, but no daily reminder.
  Interventions: Other: Educational materials

INTERVENTIONS:
Other: Daily reminders of taking medications — Reminders. Participants will receive medication-taking reminders from the researcher. These reminders are sent through the mobile application-BB Reminder on an unencrypted external device (a phone borrowed from Duke University School of Nursing and is used specifically for this study by the researcher). BB Reminder has the function that after inputting a patient's phone number and prescriptions, participants can receive reminders through text messages of the name, dosage, function, and administration route for every dose of his/her medications. The daily reminders will be sent to participants 15 minutes before every dose of their medications.
  Arms: Mobile App Group
Other: Educational materials — Educational materials. Participants will receive educational materials from the researcher. These educational materials will be sent through the mobile application-WeChat. The educational materials include short articles (< 500 words) and/or pictures. They will be retrieved from the Chinese Cardiovascular Disease-Prevention Information Website (www.healthyheart-china.com), which is governed by the Chinese Ministry of Health. The validity of information from it is guaranteed. The retrieved educational materials will be screened by the cardiologist, the head nurse, and the researcher, before sending to participants. The educational materials will be sent to participants every other day at any time during 8 am and 10 pm.

SUMMARY:
This study evaluates the feasibility and acceptability of using mobile applications to improve medication adherence. Participants in the experimental group will receive educational materials and daily reminders through mobile applications. While, participants in the control group will receive only educational materials. After the intervention, interviews will be conducted among participants through phone calls.

DETAILED DESCRIPTION:
The purpose of this study is to improve medication adherence for Chinese patients with coronary heart disease (CHD) by using mobile applications. An exploratory randomized controlled trial (RCT, N=49) and interviews (n=15) will be included in this pilot study. The RCT will compare the effects of the medication adherence (MA, n=24) intervention and control condition (n=25) on the MA score (percent of prescribed antihypertensive drugs taken), and health outcomes (SBP and DBP obtained) of patients. The health outcomes will be assessed at enrollment and every three days after the intervention begins for thirty days. Feasibility will be determined by the number of patients enrolled, and retention (percent of patients who complete the study). Acceptability (read daily reminders and educational materials via mobile applications) will be evaluated through focus group interviews. All analyses will be performed using SAS 9.3 (Cary, NC). The potential risks of this study are minimal.

ELIGIBILITY:
Inclusion criteria for participants are:

* having a medical diagnosis of CHD
* being eighteen years old or older
* having an antihypertensive medication regimen that lasts for forty-nine days or more at the enrollment
* being able to read messages through mobile phone
* having a mobile phone which can receive messages from WeChat, and can receive daily reminders from BB Reminder
* having no obvious cognitive impairment
* patients with comorbidities can be included in the study, but during the study, antihypertensive medications are their only prescribed medications (this will be screened by the cardiologist).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-07-11; Primary Completion 2016-09-19 (Actual); Study Completion 2016-11-12 (Actual)

PRIMARY OUTCOMES:
Change in medication adherence score | baseline, day 3, day 6, day 9, day 12, day 15, day 18, day 21, day 24, day 27, day 30.
  Percent of prescribed antihypertensive drugs taken during the past three days.
Change in systolic blood pressure (SBP) | baseline, day 3, day 6, day 9, day 12, day 15, day 18, day 21, day 24, day 27, day 30.
Change in diastolic blood pressure (DBP) | baseline, day 3, day 6, day 9, day 12, day 15, day 18, day 21, day 24, day 27, day 30.

SECONDARY OUTCOMES:
Feasibility as measured by patient enrollment | approximately seven weeks
  Feasibility will be determined by the number of patients enrolled, and retention (percent of patients who complete the study).
Feasibility as measured by patient retention | approximately seven weeks
  Feasibility will be determined by retention (percent of patients who complete the study)
Acceptability as measured by patient interviews | approximately seven weeks
  Acceptability (read daily reminders and educational materials via mobile applications) will be evaluated through interviews.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ni Z, Wu B, Yang Q, Yan LL, Liu C, Shaw RJ. An mHealth Intervention to Improve Medication Adherence and Health Outcomes Among Patients With Coronary Heart Disease: Randomized Controlled Trial. J Med Internet Res. 2022 Mar 9;24(3):e27202. doi: 10.2196/27202. PMID 35262490